CLINICAL TRIAL: NCT00890071
Title: Brachial Artery Peak Velocity Variation to Predict Fluid Responsiveness in Mechanically Ventilated Patients
Brief Title: Brachial Artery Peak Velocity Variation to Predict Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Hospital del SAS de Jerez (Other)
Responsible Party: Manuel Ignacio Monge García, Hospital del SAS de Jerez
Other Study IDs: UIE-SCCU-200902
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Hypotension; Shock
Keywords: Fluid responsiveness; Ultrasound; Cardiac output
MeSH Terms: conditions — Hypotension; Shock | interventions — Hypodermoclysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute circulatory failure: Patients for whom the decision to give fluids was taken because the presence of one or more clinical signs of acute circulatory failure.
  Interventions: Other: Fluid administration

INTERVENTIONS:
Other: Fluid administration — 500 ml of synthetic colloid (Voluven®, hydroxyethylstarch 6%; Fresenius, Bad Homburg, Germany) infused over 30 minutes

SUMMARY:
The investigators designed this study to determine the predictive value for predicting fluid responsiveness of noninvasive evaluation of respiratory variation of peak velocity in brachial artery, in mechanically ventilated patients with acute circulatory failure.

DETAILED DESCRIPTION:
Predicting the hemodynamic response to fluid administration (or fluid responsiveness) in critical ill patients is still a matter of concern, since fluid overload could worse the clinical situation of these patients. Parameters of fluid responsiveness usually require an invasive monitoring (like arterial pulse pressure variation).

We hypothesize that noninvasive evaluation of respiratory variation of peak velocity in brachial artery using Doppler ultrasound could provide a feasible estimation on fluid responsiveness in mechanically ventilated patients with acute circulatory failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with controlled mechanical ventilation, equipped with an indwelling radial artery catheter and for whom the decision to give fluids will be taken because the presence of one or more clinical signs of acute circulatory failure:

  * systolic blood pressure <90 mmHg (or a decrease >50 mmHg in previously hypertensive patients)
  * the need of vasopressor drugs
  * oliguria (urine output <0.5 ml/kg/min for at least 2 h)
  * tachycardia
  * delayed capillary refilling
  * the presence of skin mottling

Exclusion Criteria:

* Contraindication for the volume administration: evidence of fluid overload and/or of hydrostatic pulmonary edema
* Patients with instable cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical ill patients with controlled mechanical ventilation and acute circulatory failure.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Predictive value of respiratory variation in brachial artery peak velocity before volume expansion assessed by ROC curve. We defined responser as patients that increased stroke volume index equal or more than 15% after fluid administration. | immediately after volume expansion

SECONDARY OUTCOMES:
Evaluate the predictive value of pulse pressure variation for predicting hemodynamic response to fluid administration, comparing with the predictive value of respiratory variation of brachial artery peak velocity. | immediately after fluid administration
Evaluate the predictive value of stroke volume variation for predicting hemodynamic response to fluid administration, comparing with the predictive value of respiratory variation of brachial artery peak velocity. | immediately after volume expansion

CONTACTS AND LOCATIONS:
Overall Officials: M. Ignacio Monge García, Principal Investigator — Hospital del SAS de Jerez
Locations (1):
- Hospital del SAS de Jerez, Jerez de la Frontera, Cádiz, Spain

REFERENCES:
- [Derived] Monge Garcia MI, Gil Cano A, Diaz Monrove JC. Brachial artery peak velocity variation to predict fluid responsiveness in mechanically ventilated patients. Crit Care. 2009;13(5):R142. doi: 10.1186/cc8027. Epub 2009 Sep 3. PMID 19728876